CLINICAL TRIAL: NCT00025480
Title: A Phase I Trial of Farnesyltransferase Inhibitor, R115777 (NSC # 702818) and Radiotherapy in Patients With Non-Small Cell Lung Cancer
Brief Title: Tipifarnib Plus Radiation Therapy After Combination Chemotherapy in Treating Patients With Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068965; UPCC-NCI-5150; NCI-5150
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2007-04

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; tipifarnib; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Drug: tipifarnib
Radiation: radiation therapy

SUMMARY:
RATIONALE: Tipifarnib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by making tumor cells more sensitive to radiation therapy. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells either by killing the cells or by stopping them from dividing and may also make tumor cells more sensitive to radiation therapy.

PURPOSE: This phase I trial is studying the side effects and best dose of tipifarnib when given together with radiation therapy after combination chemotherapy in treating patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of tipifarnib given concurrently with radiotherapy after induction chemotherapy comprising paclitaxel and carboplatin and followed by maintenance therapy with tipifarnib in patients with stage IIIA or IIIB non-small cell lung cancer.
* Determine the tumor response at 3 months in patients treated with this regimen.

OUTLINE: This is multicenter, dose-escalation study of tipifarnib.

Patients receive induction chemotherapy comprising carboplatin IV over 30 minutes on day 1 and paclitaxel IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for 2 courses.

Beginning 4-6 weeks after the completion of induction chemotherapy, patients receive oral tipifarnib twice daily for 7 weeks. Patients undergo radiotherapy once daily 5 days a week for 7 weeks beginning 3 days after the start of tipifarnib. After completion of radiotherapy, patients receive oral tipifarnib twice daily for 4 days and then once daily for 4 days.

Cohorts of 3-6 patients receive escalating doses of tipifarnib while receiving radiotherapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Beginning 4-6 weeks after the completion of radiotherapy and tipifarnib, patients receive maintenance therapy comprising oral tipifarnib twice daily on days 1-21. Maintenance therapy repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3, 6, and 12 months.

PROJECTED ACCRUAL: Approximately 9-12 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Locally advanced (stage IIIA or IIIB) disease requiring radiotherapy
* No malignant pleural effusion

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* No grade 2 or greater elevation of liver function tests

Renal:

* Creatinine no greater than 1.5 times normal

Pulmonary:

* FEV_1 at least 600 cc

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No grade 3 or 4 peripheral neuropathy
* No known allergy to imidazole drugs (e.g., ketoconazole, miconazole, econazole, or terconazole)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Up to 2 prior or concurrent carboplatin and paclitaxel chemotherapy regimens allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior thoracic radiotherapy

Surgery:

* At least 3 weeks since prior exploratory thoracotomy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2001-08

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Michael Hahn, MD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States